CLINICAL TRIAL: NCT02074449
Title: Comprehensive Characterization Of Right Ventricular Performance And Afterload In Patients With Pulmonary Arterial Hypertension Undergoing Initiation And Rapid Dose Escalation Of Treprostinil
Brief Title: Study Of Right Ventricular Performance In PAH Patients Treated With Rapid Dose Treprostinil (Remodulin)
Acronym: ISS
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ISS
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2014-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Right Ventricular Performance; Treprostinil; Remodulin
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with pulmonary arterial hypertension (PAH) are at much higher risk of death if the RV (right ventricle) is weak. The purpose of this study is to get a better understanding of the factors that determine RV adaptation and how the RV compensates on therapy. The investigator is also interested in how Remodulin (treprostinil) infused over a short period (approximately 48-72 hours) affects the patient's quality of life, medical care, and personal health behaviors.

Treprostinil, also known as Remodulin, has been approved by the US Food and Drug Administration for use in the treatment of PAH. The investigator has been treating patients with Remodulin by rapid infusion (over 48 hours) for over 6 years. The investigator would like to establish this practice as safe and effective for the benefit of other centers that treat PAH.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically suspected World Health Organization (WHO) group I PAH
* Patients with New York Heart Association/WHO functional class II-IV
* Patients with mean pulmonary artery pressure >25 mmHg, pulmonary capillary wedge pressure </=15 mmHg, and pulmonary vascular resistance >3 wood units
* Age >18 and <80
* No evidence of active ischemic heart disease

Exclusion Criteria:

* Left ventricular ejection fraction <50%
* Patients with significant restrictive lung disease (FVC <60% predicted) and/or significant obstructive lung disease (FEV1 <55% predicted) within 1 year of enrollment if pulmonary function testing is available
* Patients with significant, investigator-determined parenchymal lung disease on chest x-ray or CT of the chest
* History of pulmonary embolism within the last three months or chronic pulmonary embolism
* Poorly interpretable grey scale echocardiographic images
* Contraindications to right heart catheterization
* Moderate-severe aortic and mitral valve abnormality
* Active or previous use of pulmonary vasoactive medication within the previous 12 weeks
* Renal failure with serum creatinine clearance <30 ml/hr
* High-probability ventilation-perfusion scan

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Pulmonary Arterial Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Measurement of change in RV coupling index on treprostinil between baseline, titration at 48-72 hours, and 3 months. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Franz Rischard, D.O., Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States